CLINICAL TRIAL: NCT03013595
Title: The Effectiveness of Managed Transition in Improving the Health and Social Outcomes for Young People Transitioning From Child to Adult Mental Health Care: the MILESTONE Study
Brief Title: The MILESTONE Study: Improving Transition From Child to Adult Mental Health Care
Acronym: MILESTONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Warwick (Other)
Collaborators: European Union (Other); IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other); King's College London (Other); University Hospital, Montpellier (Other); Yulius (Unknown); University of Ulm (Other); KU Leuven (Other); University College Dublin (Other); Clinical Hospital Center, Split (Other); HealthTracker Ltd, UK (Unknown); Erasmus Medical Center (Other); Concentris research management gmbh (Unknown)
Responsible Party: Principal Investigator, Swaran Singh, Professor, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: REC15/WM/0052; ISRCTN83240263 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2016-12-28; First posted 2017-01-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Mental Health Impairment; Mental Health Disorder
Keywords: Mental health; Youth mental health; Adolescent; Health services; Transition; Longitudinal cohort study; Cluster randomised controlled trial; Young adult
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRAM feedback (Experimental): 1. The completion of the "Transition Readiness and Appropriateness Measure" (TRAM, a standardized structured assessment ) prior to the transition boundary by the child and adolescent mental health service (CAMHS) clinician, young person and parent/carer.
  2. Feedback of TRAM findings to the CAMHS clinician to support decisions made regarding transition, communication with stakeholders and the transition process. Clinicians will be expected to communicate the findings to the young person and parent/carer, and, if a referral is made, to send the TRAM feedback to the adult clinician along with the referral letter.
  3. The clinicians will also receive information prior to recruitment begin on the use of TRAM and the way in which it fits in with optimal transition.
  Interventions: Behavioral: TRAM feedback
- Usual care (No Intervention): Patients, parent/carers and clinicians in the control arm will complete the TRAM prior to the transition boundary, but the clinicians won't receive any feedback from it nor any information on the benefits of using the decision support tool.

INTERVENTIONS:
Behavioral: TRAM feedback
  Other Names: Managed transition
  Arms: TRAM feedback

SUMMARY:
This study evaluates the longitudinal health and social outcomes of adolescent mental health service users who are at the transition boundary of their child and adolescent mental health service, and whether the implementation of a model of managed transition at the service boundary benefits them, as compared to usual care.

DETAILED DESCRIPTION:
The MILESTONE study focuses on the period when young people attending a children and adolescents mental health service (CAMHS) need to move on, or "transition", to an adult mental health service (AMHS), if they still require care or treatment. We know from other research that this transition is not always properly managed and that improving the transition process can have a positive impact on the health and well-being of young people in this position. We want to evaluate what impact the different transition experiences have on young people's health and well-being, and whether the process of Managed Transition has any benefits as compared to usual care.

The MILESTONE study is run in eight European countries (UK, Ireland, Belgium, Holland, France, Germany, Italy and Croatia). CAMHS in the study regions are selected to provide the young people in their care that are reaching transition age either usual care or a novel service called "Managed Transition", which includes the use of a new decision support tool, the Transition Readiness and Appropriateness Measure (TRAM). This should help with decision making and enable better transitions by identifying cases for whom transition from CAMHS to AMHS is advisable and appropriate, or who can be safely discharged or referred to a community based service. CAMHS are randomly assigned to provide the intervention of Managed Transition or usual care. The health and well-being of the young people attending these services is assessed at the start of the study and then followed-up for 24 months to see whether they transition to AMHS or are discharged or referred to some other service.

ELIGIBILITY:
Inclusion Criteria:

* Young person inclusion:

  1. Provides valid written informed consent, or assent, if below the legal age of consent
  2. If age is within one year of reaching the transition boundary of their CAMHS during the trial recruitment period, and, in exceptional cases, not more than 3 months older than the transition boundary, if a decision about transition has not yet been made
  3. Has a mental disorder defined by DSM-IV-TR, DSM-5 or ICD 10/11, or is under the regular care of CAMHS (if not yet diagnosed)
  4. Has an IQ ≥ 70 as ascertained by previous standardised assessment or diagnosed by clinician, or no indication of intellectual impairment

Exclusion Criteria:

* 1. Does not provide valid written informed consent, or assent, if below the legal age of consent 2. Is younger than a year before the transition boundary of their CAMHS 3. Has intellectual impairment (IQ <70) as ascertained by previous standardised assessment or diagnosed by clinician (if no data on intellectual functioning are available [because it has never been assessed] then care coordinators will be asked to make a clinical judgement on intellectual impairment before baseline assessment takes place) 4. If not able to (or expected not to be able to) complete the questionnaires due to severe physical disabilities or language problems, even with assistance from family members or research assistant 5. Service user in a secure forensic institution

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mental health status (need for care) as measured by Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA - clinician version) at 15 months | 15 months
  The measure will be completed by a trained MILESTONE research assistant taking into account all available sources of information (including the young person, parent/carer, relevant clinician and the medical records) to ensure accuracy of data.

SECONDARY OUTCOMES:
Self-rated (i.e. completed by young person) mental health status (need for care) on Health of the Nation Outcome Scale for Children and Adolescents (HONOSCA) | Baseline, 9, 15, and 24 months
Transition outcome assessed by the Transition Related Outcome Measure (TROM) questionnaire | Baseline, 9, 15, and 24 months
  The TROM is a questionnaire completed by the young person, parent/carer and clinician
Emotional and behavioural problems assessed by the Achenbach System of Empirically Based Assessment (ASEBA) Youth Self Report (YSR)/Adult Self Report (ASR) questionnaires (young person) | Baseline, 9, 15, and 24 months
  YSR is completed by young people aged 17 years or less; ASR by those 18 years or over
Emotional and behavioural problems assessed by the Achenbach System of Empirically Based Assessment (ASEBA) Child Behavior Checklist (CBCL) or Adult Behavior Checklist (ABCL) questionnaires (parent/carer) | Baseline, 9, 15, and 24 months
  Parent/carer completes CBCL if young person is 17 years or less; ABCL if young person is 18 years or over
Illness severity assessed by Clinical Global Impression Severity (CGIS) scale (CGIseverity) | Baseline, 9, 15, and 24 months
Quality of life assessed by World Health Organisation Quality of Life Assessment (WHOQOLBREF) | Baseline, 15, and 24 months
Independent behaviour assessed by Independent Behaviour During Consultation Scale (IBDCS) | Baseline, 9, 15, and 24 months, if young person is a current service user
Illness perception assessed by the Brief Illness Perception Questionnaire (BIPQ) | Baseline and 24 months
Barriers to care assessed by Barriers to Care (BtC) checklist | 9, 15, and 24 months, if young person is no longer a service user
Transition experience and readiness assessed by On Your Own Feet - Transition Experience Scale (OYOF-TES) | at 9, 15 or 24 months, completed only once at the first assessment after transition
Adult functioning assessed by Specific Levels of Functioning Scale (SLOF) | Baseline and 24 months
Quality Adjusted Life Years (QALYs) assessed by EuroQol generic quality of life questionnaire (EQ-5D-5L) | Baseline, 9, 15, and 24 months
Service use assessed by a MILESTONE specific Client Service Receipt Inventory (CSRI) | Baseline, 9, 15, and 24 months
Mental health status as measured by Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA - clinician version) | Baseline, 9 months, 24 months
  The measure will be completed by a trained MILESTONE research assistant taking into account all available sources of information (including the young person, parent/carer, relevant clinician and the medical records) to ensure accuracy of data.

CONTACTS AND LOCATIONS:
Overall Officials: Swaran P Singh, MD, DM, Principal Investigator — Warwick Medical School, University of Warwick, UK
Locations (10):
- Katholieke Universiteit Leuven, Leuven, Belgium
- University Hospital Split, Split, Croatia
- CHRU Montpellier-St Eloi hospital, Montpellier, France
- University of Ulm, Ulm, Germany
- University College Dublin, Dublin, Ireland
- IRCCS Fatebenefratelli, Brescia, Italy
- Netherlands (2):
  - Yulius Academy, Barendrecht
  - Erasmus Medical Centre, Rotterdam
- United Kingdom (2):
  - Warwick Medical School, University of Warwick, Coventry
  - King's College London, London

REFERENCES:
- [Derived] Marcolini F, Magno M, Leone S, Martella D, Leucci AC, Atti AR, Cortese S, De Ronchi D, Dieleman G, Franic T, Gerritsen S, Maras A, McNicholas F, Purper-Ouakil D, Santosh P, Schulze UME, Street C, Singh S, Tremmery S, Tuomainen H, van Bodegom LS, Wolke D, de Girolamo G; MILESTONE Consortium. Bridging Perspectives: Clinician-Adolescent Agreement on Psychopathological Severity in the European MILESTONE Cohort. J Clin Psychol. 2025 Nov 30. doi: 10.1002/jclp.70073. Online ahead of print. PMID 41319312
- [Derived] Magno M, Martella D, Leone S, Allibrio G, Bertani A, Caselani E, Conti P, Cortese S, Dieleman G, Franic T, Gerritsen S, Maffezzoni D, Margari F, Martinelli O, McNicholas F, Micciolo R, Nacinovich R, Purper Ouakil D, Pastore A, Rinaldi F, Santosh P, Scocco P, Schulze U, Singh S, Squarcia A, Stagi P, Street C, Toffol E, Tuomainen H, van Bodegom LS, Vicari S, de Girolamo G; on behalf the MILESTONE Consortium. Mental health trajectories of adolescents treated with psychotropic medications: insights from the european milestone study. Mol Psychiatry. 2026 Jan;31(1):94-103. doi: 10.1038/s41380-025-03307-3. Epub 2025 Oct 17. PMID 41107439
- [Derived] Gerritsen SE, Maras A, van Bodegom LS, Overbeek MM, Verhulst FC, Wolke D, Appleton R, Bertani A, Cataldo MG, Conti P, Da Fonseca D, Davidovic N, Dodig-Curkovic K, Ferrari C, Fiori F, Franic T, Gatherer C, De Girolamo G, Heaney N, Hendrickx G, Kolozsvari A, Levi FM, Lievesley K, Madan J, Martinelli O, Mastroianni M, Maurice V, McNicholas F, O'Hara L, Paul M, Purper-Ouakil D, de Roeck V, Russet F, Saam MC, Sagar-Ouriaghli I, Santosh PJ, Sartor A, Schandrin A, Schulze UME, Signorini G, Singh SP, Singh J, Street C, Tah P, Tanase E, Tremmery S, Tuffrey A, Tuomainen H, van Amelsvoort TAMJ, Wilson A, Walker L, Dieleman GC; Milestone consortium. Cohort profile: demographic and clinical characteristics of the MILESTONE longitudinal cohort of young people approaching the upper age limit of their child mental health care service in Europe. BMJ Open. 2021 Dec 16;11(12):e053373. doi: 10.1136/bmjopen-2021-053373. PMID 34916319
- [Derived] Santosh P, Singh J, Adams L, Mastroianni M, Heaney N, Lievesley K, Sagar-Ouriaghli I, Allibrio G, Appleton R, Davidovic N, de Girolamo G, Dieleman G, Dodig-Curkovic K, Franic T, Gatherer C, Gerritsen S, Gheza E, Madan J, Manenti L, Maras A, Margari F, McNicholas F, Pastore A, Paul M, Purper-Ouakil D, Rinaldi F, Sakar V, Schulze U, Signorini G, Street C, Tah P, Tremmery S, Tuffrey A, Tuomainen H, Verhulst F, Warwick J, Wilson A, Wolke D, Fiori F, Singh S; MILESTONE Consortium. Validation of the Transition Readiness and Appropriateness Measure (TRAM) for the Managing the Link and Strengthening Transition from Child to Adult Mental Healthcare in Europe (MILESTONE) study. BMJ Open. 2020 Jun 23;10(6):e033324. doi: 10.1136/bmjopen-2019-033324. PMID 32580979
- [Derived] Santosh P, Adams L, Fiori F, Davidovic N, de Girolamo G, Dieleman GC, Franic T, Heaney N, Lievesley K, Madan J, Maras A, Mastroianni M, McNicholas F, Paul M, Purper-Ouakil D, Sagar-Ouriaghli I, Schulze U, Signorini G, Street C, Tah P, Tremmery S, Tuomainen H, Verhulst FC, Warwick J, Wolke D, Singh J, Singh SP; MILESTONE Consortium. Protocol for the development and validation procedure of the managing the link and strengthening transition from child to adult mental health care (MILESTONE) suite of measures. BMC Pediatr. 2020 Apr 16;20(1):167. doi: 10.1186/s12887-020-02079-9. PMID 32299401
- [Derived] Tuomainen H, Schulze U, Warwick J, Paul M, Dieleman GC, Franic T, Madan J, Maras A, McNicholas F, Purper-Ouakil D, Santosh P, Signorini G, Street C, Tremmery S, Verhulst FC, Wolke D, Singh SP; MILESTONE consortium. Managing the link and strengthening transition from child to adult mental health Care in Europe (MILESTONE): background, rationale and methodology. BMC Psychiatry. 2018 Jun 4;18(1):167. doi: 10.1186/s12888-018-1758-z. PMID 29866202
- [Derived] Singh SP, Tuomainen H, Girolamo G, Maras A, Santosh P, McNicholas F, Schulze U, Purper-Ouakil D, Tremmery S, Franic T, Madan J, Paul M, Verhulst FC, Dieleman GC, Warwick J, Wolke D, Street C, Daffern C, Tah P, Griffin J, Canaway A, Signorini G, Gerritsen S, Adams L, O'Hara L, Aslan S, Russet F, Davidovic N, Tuffrey A, Wilson A, Gatherer C, Walker L; MILESTONE Consortium. Protocol for a cohort study of adolescent mental health service users with a nested cluster randomised controlled trial to assess the clinical and cost-effectiveness of managed transition in improving transitions from child to adult mental health services (the MILESTONE study). BMJ Open. 2017 Oct 16;7(10):e016055. doi: 10.1136/bmjopen-2017-016055. PMID 29042376